CLINICAL TRIAL: NCT02106104
Title: A Phase 4, Monocenter, Randomized, Double-blind, Comparator-controlled, Parallel-group, Mechanistic Intervention Trial to Assess the Effect of 8-week Treatment With the Dipeptidyl Peptidase-4 Inhibitor (DPP-4i) Linagliptin Versus the Sulfonylurea (SU) Derivative Glimepiride on Renal Physiology and Biomarkers in Metformin-treated Patients With Type 2 Diabetes Mellitus (T2DM)
Brief Title: Renal Effects of DPP-4 Inhibitor Linagliptin in Type 2 Diabetes
Acronym: RENALIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, M.H.H. Kramer, MD PhD, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DC2013RENALIS; U1111-1143-9518 (Other: Universal Trial Number); 2013-002493-47 (EudraCT Number); NL47157.029.13 (Registry Identifier: CCMO)
Record Dates: First submitted 2014-03-28; First posted 2014-04-08 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes mellitus; Diabetic kidney disease; Diabetic nephropathy; Renoprotection; DPP-4 inhibitors; Linagliptin; SU derivatives; Glimepiride
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies | interventions — Linagliptin; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Linagliptin 5 mg QD (N=24) (Experimental): Linagliptin 5 mg will be taken orally, once daily for 8 weeks
  Interventions: Drug: Linagliptin 5 mg QD (N=24)
- Glimepiride 1 mg QD (N=24) (Active Comparator): Glimepiride 1 mg will be taken orally, once daily for 8 weeks
  Interventions: Drug: Glimepiride 1 mg QD (N=24)

INTERVENTIONS:
Drug: Linagliptin 5 mg QD (N=24) — Linagliptin 5 mg will be taken orally, once daily for 8 weeks
  Other Names: Trajenta
  Arms: Linagliptin 5 mg QD (N=24)
Drug: Glimepiride 1 mg QD (N=24) — Glimepiride 1 mg will be taken orally, once daily for 8 weeks
  Other Names: Amaryl
  Arms: Glimepiride 1 mg QD (N=24)

SUMMARY:
The aim of this study is to detail the (mechanisms underlying the) actions of the DPP-4 inhibitor linagliptin on the renal system in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Based on preclinical and small-sized studies in non-diabetic individuals, incretin-based therapies, i.e. glucagon-like peptide (GLP)-1 receptor agonists and dipeptidyl peptidase-4 inhibitors (DPP-4i), may hold promise in preventing the onset and progression of diabetic kidney disease. However, the potential renoprotective effects of these agents, that are believed to be effectuated "beyond glucose control", have not been sufficiently detailed in human diabetes.

Therefore, the present study aims to explore the mechanistic and clinical effects of DPP-4i on fasting and postprandial renal physiology and biomarkers in patients with type 2 diabetes.

Forty-eight patients with type 2 diabetes will undergo an eight week intervention with linagliptin or glimepiride in order to assess changes in the outcome parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes (HbA1c: 6.5-9.0% DCCT or 48-75 mmol/mol IFCC)
* Metformin monotherapy; using a stable dose for at least 3 months prior to inclusion
* Both genders (females must be post-menopausal)
* Caucasian
* Age: 35-75 years
* Body Mass Index: >25 kg/m2
* All patients with previously diagnosed hypertension should use a RAS-interfering agent (angiotensin converting enzyme inhibitor/angiotensin II receptor blocker) for at least 3 months

Exclusion Criteria:

* Current / chronic use of the following medication: thiazolidinediones, insulin, glucocorticoids, immune suppressants, antimicrobial agents or chemotherapeutics. Subjects on diuretics will only be excluded when these drugs (e.g. hydrochlorothiazide) cannot be stopped for the duration of the study
* Chronic use of NSAIDs will not be allowed, unless used as incidental medication (1-2 tablets) for non-chronic indications. However, no such drugs can be taken within a time-frame of 2 weeks prior to renal-testing
* Pregnancy
* Frequent occurrence of (confirmed) hypoglycemia (plasma glucose <3.9 mmol/L)
* Estimated Glomerular Filtration Rate < 60 mL/min/1.73m2 (determined by the Modification of Diet in Renal Disease (MDRD) study equation)
* Current urinary tract infection and active nephritis
* Recent (<6 months) history of cardiovascular disease, including: acute coronary syndrome, chronic heart failure (New York Heart Association grade II-IV), stroke, transient ischemic neurologic disorder
* Complaints compatible with or established gastroparesis and/or neurogenic bladder
* Active liver disease
* History of or actual pancreatic disease
* History of or actual malignancy (except for basal cell carcinoma)
* History of or actual severe mental disease
* Substance abuse (alcohol: defined as >4 units/day; smoking/nicotine: defined as daily smoking/use)
* Allergy to any of the agents used in the study
* Inability to understand the study protocol or give informed consent

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Changes from baseline following 8-week treatment with linagliptin vs glimepiride on fasting and postprandial renal hemodynamics, measured as GFR / ERPF (determined by inulin/para-aminohippuric-acid clearance) | 8 weeks

SECONDARY OUTCOMES:
Renal tubular function | 8 weeks
Renal damage, measured by urine biomarkers | 8 weeks
Blood Pressure and Heart Rate | 8 weeks

OTHER OUTCOMES:
Body anthropometrics: body weight, height, body mass index, waist circumference | 8 weeks
Body fat content | 8 weeks
Systemic hemodynamic variables (blood pressure, heart rate, stroke volume, cardiac output/-index, total systemic vascular resistance) | 8 weeks
  Derived from non-invasive beat-to-beat finger blood pressure measurements
Cardiac autonomic nervous system function | 8 weeks
Microvascular function | 8 weeks
Arterial stiffness | 8 weeks
Glycemic variables | 8 weeks
  Glycated hemoglobin (HbA1c) and fasting glucose
Lipid spectrum | 8 weeks
DPP4- and ACE activity | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kramer, MD PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Muskiet MHA, Tonneijck L, Smits MM, Kramer MHH, Ouwens DM, Hartmann B, Holst JJ, Touw DJ, Danser AHJ, Joles JA, van Raalte DH. Effects of DPP-4 Inhibitor Linagliptin Versus Sulfonylurea Glimepiride as Add-on to Metformin on Renal Physiology in Overweight Patients With Type 2 Diabetes (RENALIS): A Randomized, Double-Blind Trial. Diabetes Care. 2020 Nov;43(11):2889-2893. doi: 10.2337/dc20-0902. Epub 2020 Sep 8. PMID 32900785